CLINICAL TRIAL: NCT02758093
Title: An RCT of Speed of Processing Training in Middle-Aged and Older Adults With HIV
Brief Title: Speed of Processing Training in Adults With HIV
Acronym: SOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Vance, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F160122002
Record Dates: First submitted 2016-03-21; First posted 2016-05-02 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: HIV; Cognition - Other; Impaired Driving

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Speed of Processing Training (10 hours) (Experimental): Participants randomized to this arm will receive 10 hours of speed of processing training; this training is designed to improve the speed/accuracy in which they identify and locate visual information using five games/exercises from the POSIT Science Speed of Processing Training. Those who receive 20 hours of speed of processing training will be compared to those participants who are randomized only to receive 10 hours speed of processing training; both of these groups will be compared to those randomized to receive only 10 hours of a computer training (Contact Control Group).
  Interventions: Behavioral: Speed of Processing Training
- Speed of Processing Training (20 hours) (Experimental): Participants randomized to this arm will receive 20 hours of speed of processing training; this training is designed to improve the speed/accuracy in which they identify and locate visual information using five games/exercises from the POSIT Science Speed of Processing Training. Those who receive 20 hours of speed of processing training will be compared to those participants who are randomized only to receive 10 hours speed of processing training; both of these groups will be compared to those randomized to receive only 10 hours of a computer training (Contact Control Group).
  Interventions: Behavioral: Speed of Processing Training
- Internet Navigational (10 hours) (Sham Comparator): In this group, participants will receive 10 hours of Internet Navigation Training. Specifically, participants will be given instructional materials and exercises on how to navigate the Internet. For more computer savvy participants, they will be directed to the Thinks.com website. Those who receive 20 hours of speed of processing training will be compared to those participants who are randomized only to receive 10 hours speed of processing training; both of these groups will be compared to those randomized to receive only 10 hours of a computer training (Contact Control Group).
  Interventions: Other: Internet Navigational

INTERVENTIONS:
Behavioral: Speed of Processing Training — These are specific computerized exercises that are designed to increase the rate in which people can process visual information.
  Other Names: Insight Software
  Arms: Speed of Processing Training (10 hours); Speed of Processing Training (20 hours)
Other: Internet Navigational — This is a sham condition in which participants will receive the same amount of social and computer contact as those randomized to receive the 10 hours of speed of processing training. In this condition, participants will learn how to do various activities on the internet.
  Other Names: Contact Control Condition
  Arms: Internet Navigational (10 hours)

SUMMARY:
As people age with HIV, the synergistic effects with normal age-related cognitive declines will accentuate and/or accelerate declines in cognitive functioning which can be detected as early in one's 40s. Although interventions are needed to protect/improve cognitive functioning, one intervention already exists to improve speed of processing. NINR/NIA (January 14, 2014) announced that Speed of Processing Training used in the ACTIVE Study (N = 2,802 community-dwelling older adults) has the ability to enable "older people to maintain their cognitive abilities as they age" even 10 years after training. As shown in the ACTIVE Study, this intervention uniquely improves driving, instrumental activities of daily living (IADL), health-related quality of life, self-rated health, internal locus of control, and protects one from depression; these represent areas of needed intervention for adults with HIV as well. In adults with HIV, previous pilot studies likewise indicate speed of processing declines are associated with poorer driving simulator performance and more self-reported at-fault automobile crashes; such speed of processing declines on driving alone represent a significant public health concern. These studies also demonstrated that Speed of Processing Training improved this cognitive ability and translated into improved performance on a timed measure of IADLs. Based on prior research, this RCT proposal consists of a pre-post two-year longitudinal experimental design whereby 264 adults with HIV, 40+ years and diagnosed with HIV-Associated Neurocognitive Disorder, will be randomly assigned to one of three training conditions: 1) 10 hours of laboratory-based Speed of Processing Training, 2) 20 hours of laboratory-based Speed of Processing Training, or 3) 10 hours of a standardized computer-contact control (sham) condition.

AIM 1: Determine whether 10 vs 20 hours of speed of processing training will improve this cognitive ability at post-test, year 1, and year 2 after baseline.

AIM 2: Determine whether 10 vs 20 hours of speed of processing training will improve everyday functioning at post-test, year 1, and year 2 after baseline.

Exploratory AIM: Determine whether improvement in speed in speed of processing and/or everyday functioning over time mediate improvement quality of life (e.g., depression, health related quality of life).

DETAILED DESCRIPTION:
SPECIFIC AIMS

This research directly meets the goals of the NIH Cognitive and Emotional Health Project and the Healthy Brain Initiative which seek to "maintain or improve the cognitive performance of all adults," especially for "populations experiencing the greatest disparities and risks in cognitive health."

Significance: Using Fascati criteria, 52% - 59% of people with HIV experience HIV-associated Neurocognitive Disorder (HAND) which affects driving safety, medication adherence, and instrumental activities of daily living (IADLs). Cognitive aging in this group represents a major concern since by 2020, 70% of adults with HIV in the United States will be 50 and older. Thus, there is a growing population that is particularly vulnerable to HAND due to the co-occurrence with aging-related cognitive impairments. In our prior study (R03MH076642-01A2) conducted in the HAART era, when comparing cognitive functioning between older and younger HIV-positive and HIV-negative adults, older adults with HIV performed the worst. In the HAART era, these cognitive impairments continue to be observed in several cognitive domains including memory, reasoning/executive functioning, and one area of particular importance - speed of processing.

Speed of processing is the rate at which cognitive functions are performed. People with HIV are vulnerable to speed of processing declines, especially as they age. Such speed of processing declines are associated with poorer driving performance, and more at-fault crashes in normal older adults, as well as middle-aged (40+) and older adults with HIV, which is a growing public health concern. In the Southern U.S., specifically in the Deep South where this study will occur, these points are highly relevant because: 1) even with speed of processing declines, adults with HIV must rely on their own driving, especially in rural areas with limited public transportation; and 2) the epicenter of HIV has emerged here in the last decade, which means many lower SES adults and/or African Americans with HIV will also have HAND or borderline HAND. Regrettably, few behavioral interventions have tried to improve cognition in this pharmacologically-burdened population; and pharmacological cognitive interventions produce adverse side effects in a population already experiencing multiple comorbidities. Fortunately, some types of computerized cognitive interventions have been shown to improve cognition without adverse side-effects. Yet, only two types of computerized cognitive interventions have been conducted in adults with HIV, with one being Speed of Processing Training.

Specific Aim 1: Determine whether 10 vs 20 hours of Speed of Processing Training will improve this cognitive ability at post-test, year 1, and year 2 after baseline. Hypothesis 1- Adults with HAND or borderline HAND will have improved speed of processing over time as they engage in more hours of training compared to those in the contact control (sham) condition.

Specific Aim 2: Determine whether 10 vs 20 hours of Speed of Processing Training will improve everyday functioning at post-test, year 1, and year 2 after baseline. Hypothesis 2- Adults with HAND or borderline HAND will have improved everyday functioning (e.g., IADLs, driving, medication adherence) over time as they engage in more hours of training compared to those in the contact control (sham) condition.

Exploratory Aim: Determine whether improvement in speed of processing and/or everyday functioning over time mediate improvement in quality of life (e.g., depression, locus of control, health-related quality of life).

Innovation: We are the first to develop Speed of Processing Training and use it with older adults and those with HIV. This non-pharmacological intervention improves the rate at which normal, community-dwelling older adults process information and has been shown to improve performance in driving, IADLs, and health-related quality of life several years after training. In prior studies, we demonstrated that after only 10 hours of Speed of Processing Training, this inexpensive intervention significantly improved speed of processing and IADLs in adults with HIV in the short-term. As part of the ACTIVE Study (N = 2,802), three types of cognitive training in 6 sites across the U.S. were compared: speed of processing, memory, and reasoning. NINR/NIA (January 14, 2014) announced that Speed of Processing Training used in the ACTIVE Study enabled "older people to maintain their cognitive abilities as they age," even 10 years after training. The ACTIVE Study also examined reasoning and memory training; however, Speed of Processing Training was uniquely found also to enhance tertiary outcomes: (1) protect against depression and (2) improve self-rated health, internal locus of control, and health-related quality of life. These tertiary/quality of life outcomes are essential areas in HIV that likewise require intervention. This RCT of 264 adults with HAND or borderline HAND will extend the ability to demonstrate that we cannot only improve speed of processing and everyday functioning in the short-term, but over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

* Since driving-related factors are being examined as one of the outcomes of the intervention, participants must be licensed drivers when entering the study.
* Men and/or women
* Must be 40+ years
* English speaking
* Have HIV-Associated Neurocognitive Disorder (HAND) or borderline HAND (defined using Frascati criteria).

Exclusion Criteria:

* Because this study is longitudinal, participants not living in stable housing (e.g., halfway house) will be excluded.
* Potential participants will be excluded if they indicate that they are planning to move outside of the Birmingham metropolitan area within the next 2 years.
* Participants with significant neuromedical co-morbidities (e.g., schizophrenia, epilepsy, bipolar disorder, multiple sclerosis, Alzheimer's disease or related dementias, mental retardation)
* Legally blind or deaf (vision confirmed at baseline)
* Currently undergoing radiation or chemotherapy
* A history of brain trauma with a loss of consciousness greater than 30 minutes
* Those who have participated in our pilot studies and were randomized to the Speed of Processing Training will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Mean Speed of Processing Measures at baseline | at baseline
  Cognitive measures of speed of processing (i.e., Useful Field of View) will be used to determine whether the training was effective.
Mean Speed of Processing Measures at 10 - 12 weeks after baseline | at 10-12 weeks after baseline
  Cognitive measures of speed of processing (i.e., Useful Field of View) will be used to determine whether the training was effective.
Mean Speed of Processing Measures at 1 year after baseline | at 1 year after baseline
  Cognitive measures of speed of processing (i.e., Useful Field of View) will be used to determine whether the training was effective.
Mean Speed of Processing Measures at 2 years after baseline | at 2 years after baseline
  Cognitive measures of speed of processing (i.e., Useful Field of View) will be used to determine whether the training was effective.

SECONDARY OUTCOMES:
Driving Simulation (a measure of everyday functioning) | Baseline (first visit), Posttest (approximately 10-12 weeks after Baseline), Year 1 (1 year after Baseline), Year 2 (2 years after Baseline)
  This driving simulator generates several outcome variables including number of crashes, number of pedestrians hit, gross reaction time, and other related driving outcomes data.
Number of vehicular crashes identified in State Crash Records for the 5 years prior to enrollment | from baseline to 5 years prior to baseline
  Driving records for participants will be pull retrospectively for the past 5 years before starting the study, and then prospectively approximately 2.5 years after Baseline (first visit) and approximately 5 years after Baseline (first visit).Documented actual at-fault crashes of the participants will be determined by pulling state driving records from the Alabama Department of Motor Vehicles.
Driving Habits Questionnaire (a measure of everyday functioning) | from baseline to 5 years prior to baseline
  This questionnaire measures self-reported data on the participants' perceived ability to drive.
Timed Instrument Activities of Daily Living (a measure of everyday functioning) | Baseline (first visit), Posttest (approximately 10-12 weeks after Baseline), Year 1 (1 year after Baseline), Year 2 (2 years after Baseline)
  This test measures the time required and the accuracy in which 5 instrumental activities of daily living (e.g., counting change) are done.
Medication Adherence (a measure of everyday functioning) | Baseline (first visit), Posttest (approximately 10-12 weeks after Baseline), Year 1 (1 year after Baseline), Year 2 (2 years after Baseline)
  This is a questionnaire that assesses how well participants take their medication as prescribed.
Number of vehicular crashes identified in State Crash Records at 2.5 years after enrollment | from baseline to 2.5 years after baseline
  Driving records for participants will be pull retrospectively for the past 5 years before starting the study, and then prospectively approximately 2.5 years after Baseline (first visit) and approximately 5 years after Baseline (first visit).Documented actual at-fault crashes of the participants will be determined by pulling state driving records from the Alabama Department of Motor Vehicles.
Number of vehicular crashes identified in State Crash Records at 5 years after enrollment | from baseline to 5 years after baseline
  Driving records for participants will be pull retrospectively for the past 5 years before starting the study, and then prospectively approximately 2.5 years after Baseline (first visit) and approximately 5 years after Baseline (first visit).Documented actual at-fault crashes of the participants will be determined by pulling state driving records from the Alabama Department of Motor Vehicles.

OTHER OUTCOMES:
Centers for Epidemiological Studies Depression Scale (a quality of life measure) | Baseline (first visit), Posttest (approximately 10-12 weeks after Baseline), Year 1 (1 year after Baseline), Year 2 (2 years after Baseline)
  This is a questionnaire that assesses how much participants identify to 20 verbal symptoms of depression.
Internal Locus of Control (a quality of life measure) | Baseline (first visit), Posttest (approximately 10-12 weeks after Baseline), Year 1 (1 year after Baseline), Year 2 (2 years after Baseline)
  This is a questionnaire that assesses the degree to which participants can exert influence over one's life.
Medical Outcomes Study Short Form (a quality of life measure) | Baseline (first visit), Posttest (approximately 10-12 weeks after Baseline), Year 1 (1 year after Baseline), Year 2 (2 years after Baseline)
  This is a questionnaire that assesses the participants' self-rated health and quality of life.
Cognitive Failures Questionnaire (a quality of life measure) | Baseline (first visit), Posttest (approximately 10-12 weeks after Baseline), Year 1 (1 year after Baseline), Year 2 (2 years after Baseline)
  This is a questionnaire that assesses what type of cognitive cognitive complaints (e.g., Do you forget where you put something like a newspaper or book?") participants experience..

CONTACTS AND LOCATIONS:
Overall Officials: David E Vance, PhD, Principal Investigator — University of Alabama at Birmingham, School of Nursing
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the cleaned electronic database available to NIMH after the study is complete.

REFERENCES:
- [Background] Vance DE, Fazeli PL, Ross LA, Wadley VG, Ball KK. Speed of processing training with middle-age and older adults with HIV: a pilot study. J Assoc Nurses AIDS Care. 2012 Nov-Dec;23(6):500-10. doi: 10.1016/j.jana.2012.01.005. Epub 2012 May 11. PMID 22579081
- [Background] Vance DE, Fazeli PL, Moneyham L, Keltner NL, Raper JL. Assessing and treating forgetfulness and cognitive problems in adults with HIV. J Assoc Nurses AIDS Care. 2013 Jan-Feb;24(1 Suppl):S40-60. doi: 10.1016/j.jana.2012.03.006. PMID 23290376
- [Background] Vance DE. Prevention, Rehabilitation, and Mitigation Strategies of Cognitive Deficits in Aging with HIV: Implications for Practice and Research. ISRN Nurs. 2013;2013:297173. doi: 10.1155/2013/297173. Epub 2013 Feb 3. PMID 23431469
- [Background] Lin F, Chen DG, Vance D, Mapstone M. Trajectories of combined laboratory- and real world-based speed of processing in community-dwelling older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):364-73. doi: 10.1093/geronb/gbs075. Epub 2012 Sep 11. PMID 22967505
- [Background] Fazeli PL, Ross LA, Vance DE, Ball K. The relationship between computer experience and computerized cognitive test performance among older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):337-46. doi: 10.1093/geronb/gbs071. Epub 2012 Aug 28. PMID 22929395
- [Background] Kaur J, Dodson JE, Steadman L, Vance DE. Predictors of improvement following speed of processing training in middle-aged and older adults with HIV: a pilot study. J Neurosci Nurs. 2014 Feb;46(1):23-33. doi: 10.1097/JNN.0000000000000034. PMID 24399164
- [Derived] Vance DE, Fazeli PL, Azuero A, Frank JS, Wadley VG, Raper JL, Pope CN, Jacob A, Ball KK. A 2-Year, Randomized, Clinical Trial Examining the Effects of Speed of Processing Cognitive Training on Quality-of-Life Indicators in Adults With HIV-Associated Neurocognitive Disorder in Birmingham, Alabama: Results of the Think Fast Study. J Assoc Nurses AIDS Care. 2024 Mar-Apr 01;35(2):104-121. doi: 10.1097/JNC.0000000000000449. Epub 2024 Jan 18. PMID 38949906
- [Derived] Vance DE, Fazeli PL, Azuero A, Frank JS, Wadley VG, Raper JL, Pope CN, Ball KK. A 2-year longitudinal randomized controlled trial examining the transfer of speed of processing training to secondary cognitive domains in middle-aged and older adults with HIV-associated neurocognitive disorder: Results of the think fast study. Clin Neuropsychol. 2024 Feb;38(2):471-492. doi: 10.1080/13854046.2023.2212867. Epub 2023 May 16. PMID 37191339
- [Derived] Waldrop D, Irwin C, Nicholson WC, Lee CA, Webel A, Fazeli PL, Vance DE. The Intersection of Cognitive Ability and HIV: A Review of the State of the Nursing Science. J Assoc Nurses AIDS Care. 2021 May-Jun 01;32(3):306-321. doi: 10.1097/JNC.0000000000000232. PMID 33449578
- [Derived] Vance DE, Robinson J, Walker TJ, Tende F, Bradley B, Diehl D, McKie P, Fazeli PL. Reactions to a Probable Diagnosis of HIV-Associated Neurocognitive Disorder: A Content Analysis. J Assoc Nurses AIDS Care. 2020 May-Jun;31(3):279-289. doi: 10.1097/JNC.0000000000000120. PMID 31436599
- [Derived] Vance DE, Cody SL, Nicholson WC, Cheatwood J, Morrison S, Fazeli PL. The Association Between Olfactory Function and Cognition in Aging African American and Caucasian Men With HIV: A Pilot Study. J Assoc Nurses AIDS Care. 2019 Sep-Oct;30(5):e144-e155. doi: 10.1097/JNC.0000000000000086. PMID 31259847
- [Derived] Vance DE, Lee L, Munoz-Moreno JA, Morrison S, Overton T, Willig A, Fazeli PL. Cognitive Reserve Over the Lifespan: Neurocognitive Implications for Aging With HIV. J Assoc Nurses AIDS Care. 2019 Sep-Oct;30(5):e109-e121. doi: 10.1097/JNC.0000000000000071. PMID 30865059
- [Derived] Vance DE, Cody SL, Nicholson C, Cheatwood J, Morrison S, Fazeli PL. Olfactory Dysfunction in Aging African American and Caucasian Men With HIV: A Pilot Study. J Assoc Nurses AIDS Care. 2022 May-Jun 01;33(3):e19-e30. doi: 10.1097/JNC.0000000000000061. PMID 30676359
- [Derived] Vance DE, Fazeli PL, Cheatwood J, Nicholson WC, Morrison SA, Moneyham LD. Computerized Cognitive Training for the Neurocognitive Complications of HIV Infection: A Systematic Review. J Assoc Nurses AIDS Care. 2019 Jan-Feb;30(1):51-72. doi: 10.1097/JNC.0000000000000030. PMID 30586083
- [Derived] Vance DE, Blake BJ, Brennan-Ing M, DeMarco RF, Fazeli PL, Relf MV. Revisiting Successful Aging With HIV Through a Revised Biopsychosocial Model: An Update of the Literature. J Assoc Nurses AIDS Care. 2019 Jan-Feb;30(1):5-14. doi: 10.1097/JNC.0000000000000029. PMID 30586079
- [Derived] Vance DE, Jensen M, Tende F, Raper JL, Morrison S, Fazeli PL. Individualized-Targeted Computerized Cognitive Training to Treat HIV-Associated Neurocognitive Disorder: An Interim Descriptive Analysis. J Assoc Nurses AIDS Care. 2018 Jul-Aug;29(4):604-611. doi: 10.1016/j.jana.2018.04.005. Epub 2018 Apr 23. No abstract available. PMID 29764716
- [Derived] Hossain S, Fazeli PL, Tende F, Bradley B, McKie P, Vance DE. The Potential of Computerized Cognitive Training on HIV-Associated Neurocognitive Disorder: A Case Comparison Study. J Assoc Nurses AIDS Care. 2017 Nov-Dec;28(6):971-976. doi: 10.1016/j.jana.2017.06.011. Epub 2017 Jun 23. No abstract available. PMID 28784586
- [Derived] Vance D, Fazeli P, Shacka J, Nicholson W, McKie P, Raper J, Azuero A, Wadley V, Ball K. Testing a Computerized Cognitive Training Protocol in Adults Aging With HIV-Associated Neurocognitive Disorders: Randomized Controlled Trial Rationale and Protocol. JMIR Res Protoc. 2017 Apr 26;6(4):e68. doi: 10.2196/resprot.6625. PMID 28446421